CLINICAL TRIAL: NCT06288334
Title: Exploration of the Optimal Dosage of Cetirizine in the Treatment of Allergic Diseases in Chinese Children
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dongyang Liu, Principal Investigator, Peking University Third Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PUTH PD_V 1.2
Record Dates: First submitted 2024-02-16; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Allergic Disease; Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric patients treated with cetirizine (Experimental): Pediatric patients who were being treated with cetirizine to fight allergic diseases.
  Interventions: Other: 1-3 Cetirizine Pharmacokinetic samples

INTERVENTIONS:
Other: 1-3 Cetirizine Pharmacokinetic samples — Limited sampling strategy was used in this study. For each child, only 1~3 blood samples were collected before and after cetirizine administration.

SUMMARY:
To obtain the pharmacokinetics of cetirizine in Chinese children with allergic disease.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent form was voluntarily signed by the legal guardians of the subjects (children aged ≥8 years should participate in the informed consent process and sign the informed consent form).
2. Pediatric patients, whether they are outpatients or inpatients, who require oral cetirizine therapy.
3. The children was clinically diagnosed with allergic diseases such as eczema, urticaria, asthma, and allergic rhinitis.
4. Pediatric patients had not taken other antiallergic drugs 72 hours before screening.

Exclusion Criteria:

1. Abnormal liver function (ALT or AST > 2 times the upper limit of normal).
2. Abnormal renal function (serum creatinine above the upper limit of normal or GFR < 10 mL/min)
3. Electrolyte abnormalities (potassium or magnesium < 0.8 times lower limit of normal, > 1.2 times upper limit of normal)
4. Children who were allergic to cetirizine or had a history of serious adverse reactions.
5. Pediatric patients with unstable vital signs.

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration | 0.5 ~ 48 hours before and after administration

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhou, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China